CLINICAL TRIAL: NCT02564393
Title: Secretion Induction of Neutrophil Extracellular Traps (NETs)in Inflammatory and Infectious Environment of Mucoviscidose
Brief Title: Induction of Neutrophilic Traps ( NETs ) by the Environment and Infectious Inflammatory Lung Cystic Fibrosis
Acronym: MucoNETs
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHAO09-PD / MucoNETs
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T: Control
- A: Adult with cystic fibrosis

SUMMARY:
The study is defined in 3 stages of in vitro assays :

Phase 1 : Secretion of NETs in response to lung disease and their secretion of factors.

This is a transversal study in which we compare :

* Producing NETs (DNA and proteases ) by neutrophils purified from sputum and blood of patients
* Producing NETs (DNA and proteases ) by purified neutrophils in the blood of patients and blood of control subjects

Phase 2: Mechanisms of activation of NETs secretory pathways . This phase will identify receptors (TLR ) involved in the secretion of NETs and analyze the involvement of dependent transduction pathways calcium and PKC . It will be performed on control blood neutrophils.

Phase 3: Analysis of cell death ( NETose )

This is a transversal study that will analyze :

the mode of cell death of neutrophils purified blood and sputum of patients and control blood neutrophils by flow cytometry and transmission electron microscopy .

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Men or women over 18
* Patients with mucoviscidose in stable condition, i.e. not having presented an acute push of bronchopulmonary attack requiring a antibiothérapie or a hospitalization for treatment of its disease during the 2 previous weeks
* Signed consent

Volunteers :

* Men or women over 18
* Without respiratory antecedent nor known respiratory pathology
* Signed consent

Exclusion Criteria:

Patients :

* In exclusion period of an other study

Volunteers :

* In exclusion period of an other study
* Antibiotic treatment and/or anti-inflammatory drug (AINS or corticoids) in the 2 weeks before inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pathophysiological study comparing a " Cystic fibrosis " group to a control group (adults)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
the DNA concentration secreted into the extracellular environment neutrophil activated | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Tours, Tours, France